CLINICAL TRIAL: NCT01878045
Title: Determinants of Diabetic Nephropathy in American Indians
Brief Title: Mechanisms of Diabetic Kidney Disease in American Indians
Status: Suspended | Type: Observational
Why Stopped: This study is on a temporary Administrative Hold pending further discussion for NIDDK and Tribal Leadership.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913151; 13-DK-N151
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-11-20

CONDITIONS: Nervous System; Diabetic Kidney Disease; Diabetes Mellitus, Type 2
Keywords: American Indians; Diabetic Nephropathy; Kidney Biopsy; Type 2 Diabetes Mellitus; Retinopathy; Natural History
MeSH Terms: conditions — Neurologic Manifestations; Diabetic Nephropathies; Diabetes Mellitus, Type 2; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- American Indians with type 2 diabetes: previously enrolled in OH95-DK-N037

SUMMARY:
Background:

- An ongoing study is looking at American Indians who have kidney problems caused by type 2 diabetes. Kidney disease due to type 2 diabetes is a major problem in American Indians. We previously found that early treatment of kidney disease with losartan was probably beneficial for reducing progression of the disease. Researchers now want to see if these benefits continue to be seen several years after the end of the treatment study.

Objectives:

- To study long-term benefit of losartan treatment for diabetic kidney disease in American Indians with type 2 diabetes.

Eligibility:

- Participants in the American Indian diabetic kidney disease study (OH95-DK-N037).

Design:

* Participants will have a physical exam and medical history before starting the study. Blood and urine samples will be collected.
* Participants will have a set of tests as part of this study. Those who have severe kidney problems, such as kidney failure, will only have a basic kidney exam with scans. The remaining participants will have a full urine collection and analysis. They will also provide a kidney biopsy.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
The purpose of this protocol is to examine the long-term impact of treatment with the angiotensin receptor blocker losartan on progression of diabetic kidney disease in American Indians with type 2 diabetes. Data from this protocol will also be used to guide the search for candidate biomarkers of diabetic end-organ damage in serum and urine and to identify mechanisms of diabetic kidney disease that may be amenable to new treatment strategies. All participants previously enrolled in a 6-year randomized clinical trial under Protocol OH95-DK-N037 and their first-degree relatives who have type 2 diabetes will be invited to participate. Participants in this protocol will undergo annual renal clearance studies to measure glomerular filtration rate and renal plasma flow, unless they have developed kidney failure. At each visit, we will also conduct tests of the peripheral and autonomic nervous system to determine the frequency, severity, and rate of progression of diabetic neuropathy in this cohort and identify linkages between diabetic kidney disease and diabetic neuropathy. We will also perform a kidney biopsy at the initial visit. In those who had a previous research kidney biopsy during the clinical trial, we will examine the extent of structural changes that occurred since their last kidney biopsy done at the end of the clinical trial. First-degree relatives and those who were enrolled in the clinical trial, but did not undergo a research kidney biopsy as part of that trial, will be invited to undergo a second kidney biopsy after 5-years of follow-up. Tissue from these biopsies will undergo morphometric examination and compartment-specific gene expression and epigenetic profiling. A small punch skin biopsy may be obtained at various times in some participants for assessment of intraepidermal nerve fiber density or for fibroblast culture. The skin biopsy for fibroblast culture will be done only once unless the culture fails, in which case the participant may be invited to undergo another biopsy. We may invite participants to undergo skin biopsy on several occasions for assessment of changes in nerve fiber density. We may also perform magnetic resonance imaging of the kidneys or the brain in some participants. Imaging of the kidneys will be done as near to the time of the kidney biopsy as possible. We many invite participants to undergo the brain imaging on 2 occasions about 3-5 years apart. Participants will be followed annually until death or development of end-stage renal disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for participation in the study, subjects must meet the following criteria:

* Previous enrollment in protocol OH95-DK-N037 or a first-degree relative of an enrollee who is aged greater than or equal to 18 years and has type 2 diabetes.
* Willingness, after receiving a thorough explanation of the study, to participate.

EXCLUSION CRITERIA:

Subjects will be excluded for the following reasons:

* Clinically significant disorders of the liver [cirrhosis, portal hypertension, hepatitis, increased bilirubin (greater than or equal to 1.5 mg/dl), cardiovascular disease (angina pectoris, history of myocardial infarction, left ventricular ejection fraction <40%, congestive heart failure of New York Heart Association Class I to IV), cerebrovascular disease, peripheral vascular disease, pulmonary diseases (asthma and restrictive or obstructive lung disease requiring therapy), renal-urinary disorders (calculi, urinary tract obstruction, glomerulonephritis, chronic infection), gastrointestinal disorders (nausea, vomiting, diarrhea or anorexia sufficient to cause weight loss or wasting), or hematocrit levels less than or equal to 30 percent in women or less than or equal to 35 percent in men.
* Renovascular or malignant hypertension; uncontrolled hypertension (systolic blood pressure greater than or equal to 160 or diastolic greater than or equal to 95 mm Hg) despite treatment with three antihypertensive drugs; or hypertension that is being treated with antihypertensive medicines and the primary care physician or the patient refuses to adopt the blood pressure treatment regimen outlined in the study protocol.
* Hematuria of unknown etiology. Prior to entry into the study, any subject with hematuria should be evaluated, the etiology established and documented, and treatment rendered as appropriate.
* Chronic debilitating disorders with or without treatment (e.g., systemic lupus erythematosus (SLE), cancer, amyloidosis, and chronic infection) that would interfere with the assessment of kidney function. Participants who develop these disorders after their original enrollment into one of our kidney studies will continue to be followed in the protocol.
* Currently receiving a drug regimen that includes: steroids, immunosuppressants, or investigational new drugs. Participants who receive these drugs following original enrollment into one of our kidney studies will continue to be followed in the protocol, unless they have known chronic significant effects on kidney morphology or a high incidence of adverse effects on kidney function, in which case they will be withdrawn from the study.
* Pregnancy. Women of childbearing potential must have a negative pregnancy test prior to entry and prior to each renal clearance study. Women who are pregnant will be offered the opportunity to participate following the conclusion of the pregnancy and those who become pregnant during the study will be able to resume the study following the conclusion of the pregnancy.
* Hypersensitivity to iodine.
* Bleeding disorders, since kidney biopsies could not be performed safely in these individuals.
* Massive obesity with body mass index greater than or equal to 45 kg/m(2). Kidney biopsies are more difficult and present greater hazards to persons with massive obesity.
* Conditions likely to interfere with informed consent or compliance with the protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in a clinical trial that is now completed and their first degree relatives with type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
End-Stage Renal Disease | Continuous surveillance performed independent of the research examinations
  Need for chronic renal replacement therapy or death attributed to kidney failure.

SECONDARY OUTCOMES:
Diabetic Neuropathy | Annually
  Neuropathy assessed by MNSI, measurements of cardiac autonomicneuropathy, and intraepidermal nerve fiber density
Diabetic Retinopathy | Anually
  Retinopathy assessed by graded retinal photographs using the Joslin Vision Network.
Cognitive function | Anually
  Cognition assessed using the NIH Toolbox.
Death | Continuous survelliance performed independently of the research examinations
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Looker, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S; RENAAL Study Investigators. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med. 2001 Sep 20;345(12):861-9. doi: 10.1056/NEJMoa011161. PMID 11565518
- [Background] Lewis EJ, Hunsicker LG, Clarke WR, Berl T, Pohl MA, Lewis JB, Ritz E, Atkins RC, Rohde R, Raz I; Collaborative Study Group. Renoprotective effect of the angiotensin-receptor antagonist irbesartan in patients with nephropathy due to type 2 diabetes. N Engl J Med. 2001 Sep 20;345(12):851-60. doi: 10.1056/NEJMoa011303. PMID 11565517
- [Background] Levey AS, Cattran D, Friedman A, Miller WG, Sedor J, Tuttle K, Kasiske B, Hostetter T. Proteinuria as a surrogate outcome in CKD: report of a scientific workshop sponsored by the National Kidney Foundation and the US Food and Drug Administration. Am J Kidney Dis. 2009 Aug;54(2):205-26. doi: 10.1053/j.ajkd.2009.04.029. Epub 2009 Jul 3. PMID 19577347